CLINICAL TRIAL: NCT05963100
Title: Clinical Study of TCR-like CAR-T Cell Targeted MSLN in the Treatment of Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yang Shen, Professor, Zhongda Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023010142
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Safety and Efficacy of TCR-like CAR-T

STUDY DESIGN:
Intervention Model Description: dose climbing test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1*10^6/kg (Experimental)
  Interventions: Biological: TCR-like CAR-T
- Experimental 1*10^7/kg (Experimental)
  Interventions: Biological: TCR-like CAR-T
- Experimental 3*10^6/kg (Experimental)
  Interventions: Biological: TCR-like CAR-T
- Experimental 2*10^7/kg (Experimental)
  Interventions: Biological: TCR-like CAR-T

INTERVENTIONS:
Biological: TCR-like CAR-T — intravenous drip of TCR-like CAR-T with indicated doses

SUMMARY:
The goal of this clinical trial is to test TCR-like CAR-T in the Treatment of MSLN positive Ovarian Cancer. The main question it aims to answer are: the safety and efficacy of TCR-like CAR-T in the Treatment of MSLN positive Ovarian Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced platinum-resistant ovarian cancer, with a positive rate of IHC mesothelin in tumor tissue ≥ 26% [Participants need to undergo fresh tumor tissue biopsy for biomarker analysis]. If biopsy is not possible, it is necessary to provide archived tumor tissue (at least 8 unstained FFPE sections) within 18 months. If there have been multiple tumor tissue collections in the past, the newly collected samples will be prioritized
* Non resectable advanced ovarian cancer that has failed standard treatment (has previously received at least one platinum containing systemic chemotherapy regimen) or lacks effective treatment methods
* At least 1 measurable lesion (according to RECIST 1.1 standard)
* ECOG score 0-1 and estimated survival greater than 3 months
* The laboratory test results should at least meet the following indicators: Lambda Left ventricular Ejection fraction ≥ 45%; Creatinine clearance rate ≥ 50mL/min; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Absolute lymphocyte count (ALC) ≥ 0.7 × 109/L; Platelet count (PLT) ≥ 100 × 109/L; Hemoglobin ≥ 90g/L; Blood oxygen saturation>91%; Total bilirubin ≤ 2 × ULN (upper limit of normal value): alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Researchers have determined that ALT and AST abnormalities caused by diseases (such as liver metastasis or bile duct obstruction) or Gilbert syndrome can be relaxed to ≤ 5 × ULN;
* The researcher determines that the subject needs to recover from all toxicity related to the previous treatment to an acceptable baseline state, or the relevant toxicity needs to return to normal or level 1 of the NCI CTCAE 5.0 scoring standard; Excluding toxicity that the researcher determines will not increase the safety risk of subsequent study drug reinfusion, such as hair loss, vitiligo, etc;
* Can understand this experiment and have signed an informed consent form.
* Venous access with venous or single blood collection

Exclusion Criteria:

* Other malignant tumors other than ovarian cancer in the first five years of screening, in addition to fully treated cervical Carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and Ductal carcinoma in situ after radical surgery;
* Hepatitis B B surface antigen (HBsAg) or hepatitis B B core antibody (HBcAb) is positive, and the detection result of hepatitis B virus (HBV) DNA titer in peripheral blood is higher than 50IU/ml or the lower limit of the quantitative detection range of the research center; Hepatitis C virus (HCV) antibody is positive and the peripheral blood HCV RNA detection result is higher than the lower limit of the quantitative detection range of the research center; People who are positive for human immunodeficiency virus (HIV) antibodies; Those who have tested positive for syphilis
* Patients with ovarian cancer metastasis to the central nervous system and/or other unstable Central nervous system disease (bleeding, active infarction, infection, etc.)
* Received attenuated live vaccine within 4 weeks before cell transfusion
* It is known that any ingredient used in the treatment of this study may cause allergic reactions
* Hypertension with poor drug control (systolic pressure>160mmHg and/or diastolic pressure>90mmHg) or cardio cerebral Vascular disease with clinical significance (such as activity), such as cerebrovascular accident (within 6 months before signing the master informed consent), myocardial infarction (within 6 months before signing the master informed consent), unstable angina pectoris, congestive heart failure classified as Grade II or above by New York Heart Association (NYHA), Severe arrhythmia cannot be controlled with medication or has potential impact on research and treatment; The electrocardiogram shows clinically significant abnormalities or an average QTcB of ≥ 450ms after 3 consecutive attempts (with an interval of at least 5 minutes)
* Concomitant with other serious organic or mental illnesses
* Suffering from systemic active infections that require treatment
* Suffering from autoimmune diseases: the history of Autoimmune disease determined by the researcher to be unsuitable for this study, such as systemic lupus erythematosus, vasculitis, and invasive lung diseases, should be excluded (except for Vitiligo subjects)
* Systematically available pine steroids (local use allowed), Hydroxycarbamide and immunomodulators (such as: α or γ Interferon, GM-CSF, mTOR inhibitor, cyclosporin, Thymosin, etc.)
* Chemotherapy was received 2 weeks before screening, immunotherapy was received within 4 weeks, radiation therapy was received 12 weeks before screening, or other anti-tumor treatment drugs had a washout period of less than 5 half-lives
* Pregnant or lactating women, and female subjects who plan to conceive within 1 year after cell transfusion
* Subjects with any coexisting medical conditions or diseases that the researcher determines may affect the conduct of this experiment
* Patients who have received other cell gene therapy products within 6 months prior to cell reinfusion and are considered unsuitable for inclusion by researchers
* The researcher determines that the patient is unable to complete all visits or procedures required by the research protocol (including the follow-up period), or has insufficient compliance to participate in this study; Or patients deemed unsuitable for inclusion by researchers
* Items included in the selection and exclusion criteria for the pre screening period audit

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of KT127 cells | up to second year
  The highest dose level (cells/kg) where ≤2/6 evaluable subjects experience protocol-defined dose-limiting toxicities (DLTs) within 14 days post-infusion, with dose escalation terminated based on pre-specified safety criteria.
Adverse events (AEs) | up to second year
  The ASTCT 2019 standard will be used to grade cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), and the CTCAE version 5.0 standard will be used to grade other adverse events. Unless otherwise specified in the protocol, all AEs that occur during the entire study period will be evaluated.

SECONDARY OUTCOMES:
objective response rate(ORR) | up to second year
  The objective response rate evaluation will be based on the researcher's evaluation of imaging, and the efficacy evaluation will refer to the evaluation criteria for solid tumors (RECIST 1.1) The objective response rate evaluation will be based on the researcher's evaluation of imaging, and the efficacy evaluation will refer to the evaluation criteria for solid tumors(RECIST 1.1)
progression-free survival(PFS) | up to second year
  Progressive free survival is the time from receiving investigational drug treatment to the onset of the first PD or death from any cause in the absence of documented PD
Overall survival(OS) | up to second year
  The total survival period is the time between receiving investigational drug treatment and subject death due to various reasons

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, PhD, Study Chair — Zhongda Hospital
Locations (1):
- Zhongda hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No